CLINICAL TRIAL: NCT00937625
Title: T-cell Based Immunotherapy for Treatment of Patients With Disseminated Melanoma.
Brief Title: T-cell Based Immunotherapy for of Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM0909
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine; Interleukin-2; fludarabine phosphate; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: cyclophosphamide, fludarabine, T-cells, Interleukin-2 — Two days of cyclophosphamide (60 mg/kg i.v.) and five days of fludarabine (25 mg/m2 i.v.). Infusion of Tumor Infiltrating Lymphocytes (10e9-10e10 cells). Followed by daily sc injections of 2 MIE Interleukin-2 for two weeks. After the first 6 patients the dose of IL-2 has been changed to an i.v. decrescendo regimen using 18 MIU/m2 infused over 6, 12 and 24 hours and then 4.5 MIU/m2 infused over 24 hours for three days.
  Other Names: Cyclophosphamide, Sendoxan®, Baxter A/S; Fludarabine, Fludara®, Bayer Shering; Interleukin-2, Proleukin®, Chiron B.V.

SUMMARY:
The aim of this study is to investigate the toxicity and clinical response of therapy with tumor infiltrating lymphocytes as treatment for advanced melanoma.

Patient will receive a single treatment consisting of conditioning chemotherapy for seven days (cyclophosphamide for two days and fludarabine for five days), intravenous infusion of high number of in vitro expanded tumor infiltrating lymphocytes followed by two weeks with daily low-dose interleukine-2. Patients will be evaluated for toxicity, tumor response, and immune response.

After the first 6 patients the treatment with IL-2 has been changed to include higher doses of IL-2 (see intervention)

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological proven skin derived progressive metastatic or locally advanced malignant melanoma. Further inclusion criteria: Performance Status 0 to 1, surgical available metastasis, at least one measurable lesion, acceptable CBC and blood chemistry results. Acceptable organ functions.

Exclusion Criteria:

* Patients with a history of any other malignancies less than five years ago. Brain metastases. Other significant illness including severe allergy, asthma, DM, angina pectoris, congestive heart failure, chronic infections, or active autoimmune disease. Treatment with immune suppressive drugs, experimental drugs, or antineoplastic drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
toxicity | week 0 to 20

SECONDARY OUTCOMES:
immune response | week 0 to 20
tumor response | week 8 and every 3rd week until progression

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Professor, MD, Study Director — Department of Oncology, Copenhagen University Hospital, Herlev, Herlev Ringvej 75, DK-2730 Herlev, Denmark; Rikke Andersen, MD, Principal Investigator — Center for Cancer Immune Therapy, department of Oncology, Herlev Hospital, Denmark
Locations (1):
- Department of Oncology, Copenhagen University Hospital, Herlev, Herlev, Denmark

REFERENCES:
- [Derived] Dolton G, Rius C, Wall A, Szomolay B, Bianchi V, Galloway SAE, Hasan MS, Morin T, Caillaud ME, Thomas HL, Theaker S, Tan LR, Fuller A, Topley K, Legut M, Attaf M, Hopkins JR, Behiry E, Zabkiewicz J, Alvares C, Lloyd A, Rogers A, Henley P, Fegan C, Ottmann O, Man S, Crowther MD, Donia M, Svane IM, Cole DK, Brown PE, Rizkallah P, Sewell AK. Targeting of multiple tumor-associated antigens by individual T cell receptors during successful cancer immunotherapy. Cell. 2023 Aug 3;186(16):3333-3349.e27. doi: 10.1016/j.cell.2023.06.020. Epub 2023 Jul 24. PMID 37490916
- [Derived] Kristensen NP, Heeke C, Tvingsholm SA, Borch A, Draghi A, Crowther MD, Carri I, Munk KK, Holm JS, Bjerregaard AM, Bentzen AK, Marquard AM, Szallasi Z, McGranahan N, Andersen R, Nielsen M, Jonsson GB, Donia M, Svane IM, Hadrup SR. Neoantigen-reactive CD8+ T cells affect clinical outcome of adoptive cell therapy with tumor-infiltrating lymphocytes in melanoma. J Clin Invest. 2022 Jan 18;132(2):e150535. doi: 10.1172/JCI150535. PMID 34813506
- [Derived] Borch TH, Andersen R, Ellebaek E, Met O, Donia M, Svane IM. Future role for adoptive T-cell therapy in checkpoint inhibitor-resistant metastatic melanoma. J Immunother Cancer. 2020 Jul;8(2):e000668. doi: 10.1136/jitc-2020-000668. PMID 32747469
- [Derived] Andersen R, Donia M, Ellebaek E, Borch TH, Kongsted P, Iversen TZ, Holmich LR, Hendel HW, Met O, Andersen MH, Thor Straten P, Svane IM. Long-Lasting Complete Responses in Patients with Metastatic Melanoma after Adoptive Cell Therapy with Tumor-Infiltrating Lymphocytes and an Attenuated IL2 Regimen. Clin Cancer Res. 2016 Aug 1;22(15):3734-45. doi: 10.1158/1078-0432.CCR-15-1879. Epub 2016 Mar 22. PMID 27006492
- [Derived] Donia M, Hansen M, Sendrup SL, Iversen TZ, Ellebaek E, Andersen MH, Straten Pt, Svane IM. Methods to improve adoptive T-cell therapy for melanoma: IFN-gamma enhances anticancer responses of cell products for infusion. J Invest Dermatol. 2013 Feb;133(2):545-52. doi: 10.1038/jid.2012.336. Epub 2012 Sep 27. PMID 23014345
- [Derived] Ellebaek E, Iversen TZ, Junker N, Donia M, Engell-Noerregaard L, Met O, Holmich LR, Andersen RS, Hadrup SR, Andersen MH, thor Straten P, Svane IM. Adoptive cell therapy with autologous tumor infiltrating lymphocytes and low-dose Interleukin-2 in metastatic melanoma patients. J Transl Med. 2012 Aug 21;10:169. doi: 10.1186/1479-5876-10-169. PMID 22909342